CLINICAL TRIAL: NCT07179900
Title: Exploration of Radiotherapy Combined With QL1706 and Bevacizumab for the Conversion Treatment of Unresectable Non-metastatic Hepatocellular Carcinoma: A Prospective, Open-label, Randomized Controlled Clinical Study
Brief Title: Radiotherapy Combined With QL1706 and Bevacizumab for Unresectable Non-metastatic Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025KY047
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy; sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy+QL1706+Bevacizumab (Experimental): After enrollment, patients first received radiotherapy (41.4 - 50.4 Gy/23 - 28 F). At 25.2 Gy/14 F of radiotherapy, the first systemic treatment was administered: QL1706 7.5 mg/kg + bevacizumab 15 mg/kg, once every 3 weeks. The second cycle of systemic treatment was initiated 7 - 14 days after the completion of radiotherapy. Within 2 weeks after the completion of 4 cycles of systemic treatment (including 1 cycle during radiotherapy and 3 cycles after radiotherapy), preoperative efficacy was evaluated based on the two primary endpoints of this study.
  Interventions: Drug: QL1706; Radiation: Radiotherapy; Drug: Bevacizumab
- Sintilimab+Bevacizumab (Other): After enrollment, patients were received 4 cycles of sintilimab 200mg and bevacizumab 15mg/kg, once every 3 weeks. The first efficacy assessment was conducted within 2 weeks after the end of the systemic treatment, based on the two primary endpoints of this study.
  Interventions: Drug: Sintilimab; Drug: Bevacizumab

INTERVENTIONS:
Drug: QL1706 — Apololitovoreli monoclonal antibody (QL1706) 7.5mg/kg intravenous infusion, once every 3 weeks
  Other Names: Iparomlimab and Tuvonralimab Injection
  Arms: Radiotherapy+QL1706+Bevacizumab
Radiation: Radiotherapy — 41.4-50.4Gy/1.8Gy/23-28F
  Arms: Radiotherapy+QL1706+Bevacizumab
Drug: Sintilimab — 200mg q3w
  Arms: Sintilimab+Bevacizumab
Drug: Bevacizumab — 15mg/kg q3w

SUMMARY:
This project is a prospective, open-label, randomized controlled clinical study. It plans to enroll 60 patients with unresectable HCC and no distant metastasis, randomly assigned to the experimental group and the control group, with 30 cases in each group. The experimental group was treated with radiotherapy combined with immunotherapy and Bevacizumab, while the control group was treated with immunotherapy and Bevacizumab. The efficacy of the patients and the conversion rate to surgery were evaluated.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old, gender not limited; PS score 0-2; Pathologically or clinically diagnosed as primary HCC and has not received other anti-HCC treatment; No history of other malignant tumors or treatment; Patients with BCLC stage B or C before treatment and no distant metastasis, and surgical assessment indicates that first-line surgical resection is not feasible; Liver function grade Child-Pugh A or B ≤ 7 points; For patients with active HBV infection, antiviral treatment should be initiated at least 7 days before treatment and they should agree to continue antiviral treatment during the study period; No severe cardiovascular or cerebrovascular diseases; Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the treatment period and 6 months after treatment; if the serum or urine pregnancy test is negative within 14 days before inclusion in the study, and the patient must be non-lactating; men should agree to take contraceptive measures during the study period and 6 months after the study; Voluntarily sign the written informed consent form and commit to comply with the protocol during the study period, including accepting treatment and scheduled visits and examinations, including follow-up; The expected survival must be at least 12 weeks.

Exclusion Criteria:

Patients who do not meet the above main inclusion criteria; Patients who refuse to sign the informed consent form; Patients with pathological types of cholangiocarcinoma, sarcomatoid hepatocellular carcinoma, mixed cell carcinoma and fibrolamellar cell carcinoma; or those with postoperative pathology suggesting metastatic cancer or primary cancer of other tissue types; Patients with portal hypertension diagnosed by preoperative enhanced abdominal CT and endoscopy, with a history of esophageal variceal bleeding, severe hypersplenism syndrome or refractory ascites; Patients diagnosed with severe active scleroderma, lupus, other rheumatic diseases or autoimmune diseases within the past 3 months before study recruitment; patients with a history of clinically severe autoimmune diseases or those requiring systemic steroids or immunosuppressants will not be allowed to participate in this study; Patients with a history of cognitive dysfunction or mental illness that affects treatment compliance; Patients whom the investigator deems unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  PR+CR
R0 resection rate | 1 year
  The proportion of patients achieving R0 resection

SECONDARY OUTCOMES:
pCR rate | 1 year
  The proportion of patients achieving pCR in postoperative pathology
Time of disease progression | 3 year
  The time from the start of treatment to disease progression (PD)
PFS | 3 year
  The time from randomization to disease progression (PD) or death from any cause
OS | 3 year
  The time from randomization to patient death due to various reasons.
The occurrence of treatment-related adverse events | 3 Year
  Treatment-related adverse events were evaluated and statistically summarized according to CTCAE version 5.0.

IPD SHARING:
Plan to Share IPD: No